CLINICAL TRIAL: NCT07283250
Title: Development and Validation of the Air Quality Awareness Scale (AQAS) for Parents of Children With Allergic Diseases: A Cross-sectional Study
Brief Title: Development and Validation of the Air Quality Awareness Scale (AQAS) for Parents
Status: Enrolling by invitation | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Hilal Gungor, Medical Doctor, Pediatric Immunology and Allergy, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 2025-654789651231
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Asthma (Diagnosis); Air Quality; Air Pollution; Rhinitis, Allergic; Health Knowledge, Attitudes, Practice; Health Belief Model; Parents
MeSH Terms: conditions — Asthma; Disease; Rhinitis, Allergic; Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents of Children with Allergic Airway Diseases: This cohort includes parents or primary caregivers of children aged 2-18 years who have been clinically diagnosed with allergic airway diseases (asthma and/or allergic rhinitis) by a pediatric allergy specialist. Participants will complete a structured questionnaire assessing their awareness, knowledge, and preventive behaviors regarding air pollution and air quality.
  Interventions: Behavioral: Air Quality Knowledge Questionnaire

INTERVENTIONS:
Behavioral: Air Quality Knowledge Questionnaire — A structured, self-administered questionnaire on air quality and pollution will be provided to all participants.
  The survey consists of a total of 23 main items and an additional demographic information section.
  The demographic section collects data on parent's age, gender, education level, occupation, and the child's age, gender, diagnosis (asthma and/or allergic rhinitis), and disease duration.
  The main questionnaire includes:
  * 5 items assessing knowledge of air pollution and air quality concepts;
  * 10 items measuring awareness of air pollution sources, health impacts, and environmental conditions;
  * 8 items evaluating attitudes and protective behaviors toward air pollution (e.g., monitoring air quality index, modifying outdoor activities, using indoor air filters).
  Responses are based on a Likert-type scale. The tool is designed to quantify parental understanding, awareness, and preventive practices related to air quality in the context of childhood allergic airway diseases.

SUMMARY:
This cross-sectional study aims to assess the level of awareness, knowledge, and preventive behaviors regarding air quality and air pollution among parents of children with physician-diagnosed allergic respiratory diseases (asthma and/or allergic rhinitis). The survey will evaluate parents' understanding of air pollution effects, sources, and protective measures, as well as sociodemographic and clinical correlates influencing awareness.

ELIGIBILITY:
Inclusion Criteria:

* Parent or primary caregiver of a child aged 2-18 years
* Child has a physician-diagnosed asthma and/or allergic rhinitis
* Able to read and understand Turkish
* Provides informed consent

Exclusion Criteria:

* Parents of children with other chronic respiratory or systemic diseases
* Parents who are healthcare professionals (to avoid bias)
* Incomplete survey responses

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of parents or primary caregivers of children aged 2 to 18 years who have been clinically diagnosed with allergic airway diseases, specifically asthma and/or allergic rhinitis, by a pediatric allergy specialist.
  Participants will be recruited from the outpatient Pediatric Allergy Clinic of a tertiary healthcare center.
  All participants must be able to read and understand Turkish and voluntarily provide written informed consent.
  The survey targets approximately 500 parents, representing diverse educational and socioeconomic backgrounds, to evaluate knowledge, awareness, and behaviors related to air quality and pollution.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Level of Parental Knowledge and Awareness About Air Quality | At baseline (single survey administration)
  The primary outcome is the overall score obtained from the Air Quality Knowledge and Behavior Questionnaire, reflecting parents' knowledge and awareness regarding air quality and air pollution.
  The composite score will be derived from the 5 knowledge and 10 awareness items, each rated on a Likert scale (e.g., 1 = strongly disagree to 5 = strongly agree).
  Higher total scores indicate greater knowledge and awareness of air pollution, its sources, and its health effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly because the dataset contains potentially identifiable information collected from a limited number of participants at a single center.
  Only aggregated, de-identified summary data will be included in publications and presentations.
  The study protocol and statistical analysis plan may be shared upon reasonable request from qualified researchers, following approval by the principal investigator and the institutional ethics committee.